CLINICAL TRIAL: NCT05729867
Title: Efficacy and Safety of a Fully Covered Self-Expandable Metal Stent for Unresectable Hepatocellular Carcinoma: A Prospective Cohort Study
Brief Title: Efficacy and Safety of a Fully Covered Self-Expandable Metal Stent for Unresectable HCC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sang Hyub Lee, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-2004-175-1119
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Malignant Biliary Obstruction; Hepatocellular Carcinoma
Keywords: Self expandable metal stent
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- fully covered self-expanable metal stent with HCC (Experimental): This prospective cohort is comprised of patients with malignant biliary obstruction caused by hepatocellular carcinoma who were treated with endoscopic biliary drainage using fully covered self expandable metal stent.
  Interventions: Procedure: Endoscpic biliary drainage using fully covered metal stent

INTERVENTIONS:
Procedure: Endoscpic biliary drainage using fully covered metal stent — After selective cannulation of the bile duct, cholangiography is obtained using contrast agent.
  A guide wire is passed through the stricture, and then fully-covered metal stent is inserted under fluoroscopy guidance during ERCP.

SUMMARY:
The effectiveness and safety of fully covered metal stent in malignant biliary obstruction caused by HCC are still unknown. These would be clarified in this prospective cohort study.

DETAILED DESCRIPTION:
In this study, endoscopic biliary drainage was performed using fully covered self-expancdable metal stent for malignant biliary obstruction caused by HCC. Main outcome is efficacy and safety of this procedure including clinical success rate, technical success rate, stent patency, stent dysfunction, and any adverse events during the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19 years or older, those who consented to the clinical research participation and signed a written consent form
* Obstructive jaundice caused by unresectable hepatocellular carcinoma

Exclusion Criteria:

* Patients who have previously undergone surgical biliary drainage
* Patients who need to remain percutaneous transhepatic biliary drainage
* Patients whose life expectancy is less than 3 months (BCLC stage D without a treatment plan for hepatocellular carcinoma)
* Patients who cannot undergo endoscopic procedure according to the judgment of the researcher

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-04-27 (Actual); Primary Completion 2024-04-26 (Estimated); Study Completion 2025-04-26 (Estimated)

PRIMARY OUTCOMES:
Clinical success rate | 1 month
  Clinical success rate is defined as a reduction of total bilirubin level above 50% or total bilirubin level less than 2 mg/dL within 1 month after the procedure. Clinical success rate of all procedures will be measured.
Technical success rate | 1 day
  Technical success is defined as whether the stent is properly inserted into the stricture site and the bile or contrast agent is drained. Technical success rate of all procedures will be measured.

SECONDARY OUTCOMES:
Stent patency duration | 1 year
  Stent patency duration is defined as number of days between immediately after procedure and occurrence of stent dysfunction.
Stent migration rate | 1 year
  Stent migration is divided in two types. Proximal dislocation is defined as the movement of the stent into the bile duct at the site of obstruction, and distal dislocation is defined as the distal displacement of the stent from the stenotic site (including cases where the stent is not observed due to self-removal). The rate of stent migration including both proximal and distal dislocation will be measured.
Stent dysfunction rate | 1 year
  The stent dysfunction includes stent migration, occlusion, jaundice after stent insertion (increased more than 2-fold based on the lowest total bilirubin level), situations requiring endoscopy or radiologic intervention. The stent dysfunction rate of all patients will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Sang Hyub Lee, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No